CLINICAL TRIAL: NCT02454491
Title: Comparison of VERapamil vs. Heparin Therapy on Procedural sUccess During Transradial Coronary Procedures (VERMUT Study)
Brief Title: Verapamil vs Heparin in Transradial Procedures
Acronym: VERMUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Assistant Professor and Interventional Cardiologist, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58
Record Dates: First submitted 2015-05-13; First posted 2015-05-27 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Heart Disease, Ischemic
Keywords: percutaneous coronary interventions; radial artery access; access site complications; verapamil; heparin
MeSH Terms: conditions — Myocardial Ischemia | interventions — Heparin; Verapamil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard of care (Active Comparator): intraradial heparin (5000 UI) immediately after a 6 F sheath insertion
  Interventions: Drug: Heparin
- experimental therapy (Experimental): intraradial verapamil (5 mg) immediately after a 6 F sheath insertion
  Interventions: Drug: Verapamil

INTERVENTIONS:
Drug: Heparin — intraradial administration of heparin 5000 ui
  Arms: standard of care
Drug: Verapamil — intraradial administration of verapamil 5 mg
  Arms: experimental therapy

SUMMARY:
Transradial approach (TRA) for cardiac catheterization and percutaneous coronary interventions (PCI) is increasingly being used worldwide. At the present is unknown the cocktail of agents necessary to minimize local access site complications. The investigators planned a prospective randomized clinical trial to test the superiority of verapamil vs. heparin in the reduction of access site related complications.

DETAILED DESCRIPTION:
Transradial approach (TRA) for cardiac catheterization and percutaneous coronary interventions (PCI) is increasingly being used worldwide in both elective and emergency procedures because it reduces net adverse clinical events, through a reduction in major bleeding and all-cause mortality, when compared to transfemoral approach. However, radial artery occlusion (RAO) after the procedure (the incidence of which varies from 1% to 10%) remains one of the major limitations of TRA.

The aim of the study is to assess the superiority of verapamil versus heparin in the access success during transradial percutaneous coronary interventions (PCI).

METHODS Patients referred to the cath-lab of the Cardiovascular Institute of the University Hospital of Ferrara, Italy, for coronary angiography were randomized in 2 groups with a computer-generated random sequence. The study is double-blind. In the first group, patients received intravenous heparin (5000 UI) immediately after a 6 F sheath insertion. In the second group, patients received Verapamil (5 mg) immediately after a 6 F sheath insertion. If after the start of the procedure a radial artery spasm (RAS) occurs, the operators can choose to use bail-out a local vasodilator therapy. After sheath removal, hemostasis was obtained using a TR band (Terumo corporation, Tokyo, Japan) with a plethysmography-guided patent hemostasis technique. Radial artery patency was evaluated at 24 hours (early RAO) and 30 days after the procedure (late RAO) by ultrasound.

The aim of the study is to demonstrate that verapamil administration is superior to heparin administration in the reduction of the combined endpoint (occurrence of radial artery occlusion (early RAO), access site complication, radial artery spasm (RAS) requiring local bailout use of vasodilatator)

RAO will be assessed by ultrasonography by independent expert reviewer blinded to randomization

The investigators defined access site complication the following items:

* local haematoma superficial <5 cm from access site;
* haematoma with moderate muscle infiltration <10 cm;
* forearm haematoma and muscular infiltration below the elbow;
* haematoma and muscular infiltration above the elbow;
* ischemic threat (compartmental syndrome);
* radial artery dissection during the procedure;

The investigators defined radial artery spasm any spasm occurring during the procedure requiring the administration of local vasodilatators to allow the procedure

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to hospital with diagnosis of acute coronary syndrome and stable coronary artery disease according current European guidelines and with clinical indication to coronary artery angiography.

* all patients receiving percutaneous coronary intervention by radial artery access as first attempt
* procedures with 6F catheter

Exclusion Criteria:

* warfarin therapy
* previous ipsilateral TRA
* lack of consent
* scleroderma
* thrombocytopenia
* or other contraindications to heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
number of participants with radial artery-related complications | 24 hours
  occurrence of early radial artery occlusion, access site complication, radial artery spasm (RAS) that requires the bailout use of vasodilatator

SECONDARY OUTCOMES:
number of participants with each radial artery-related complication | 24 hours
  occurrence of each singular component of primary endpoint
late radial artery occlusion | 30 days
  occurrence of radial artery occlusion (late RAO)
reopening early RAO | 30 days
  reopening of the closed radial at 24 hours.
patient's satisfaction | 24 hours
  assessment with questionnaires of the pain and satisfaction of patients
long term patient's satisfaction | 30 days
  assessment with questionnaires of the pain and satisfaction of patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy